CLINICAL TRIAL: NCT03042221
Title: Early Rebiopsy to Identify Mechanisms and Biomarkers of Tumor Cell Survival Following Systemic Therapy for Lung Cancer
Brief Title: Early Rebiopsy to Identify Biomarkers of Tumor Cell Survival Following EGFR, ALK, ROS1 or BRAF TKI Therapy
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2316.cc
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Carcinoma of Lung, TNM Stage 4; Non-Small Cell Lung Cancer; EGFR Gene Mutation; ALK Gene Mutation; ROSE Cluster 1; BRAF V600E
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A comparison of baseline tumor characteristics in oncogene-driven cancers to tumor characteristics after early response to Tyrosine Kinase Inhibitor (TKI) targeted treatment will allow identification of early adaptive mechanisms of cell survival. This will facilitate targeting and termination of these survival/ resistance pathways before they develop with rational combinations of therapeutic agents to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

Targetable Oncogene - Biopsy Cohort (includes blood draw)

1. Carry a diagnosis of locally advanced or stage IV NSCLC responsive to targeted therapies (per current NCCN guidelines)
2. Aged 18 years or older
3. ECOG 0-2
4. Have a histologically confirmed diagnosis of NSCLC harboring an activating mutation responsive to targeted therapy (per NCCN guidelines)
5. No prior systemic therapy for locally advanced or metastatic disease.
6. Planned treatment with targeted therapy specific to the oncogene driver mutation.
7. Patients must have at least one site of measurable disease ≥ 2cm.
8. Primary disease site or site of metastatic disease must be amenable to biopsy.
9. Patients must have the ability to understand and willingness to sign an informed consent document.

Targetable Oncogene - Blood Draw Only Cohort

1. Carry a diagnosis of locally advanced or stage IV NSCLC responsive to targeted therapy (per NCCN guidelines)
2. Aged 18 years or older
3. ECOG 0-2
4. Have a histologically confirmed diagnosis of NSCLC harboring an activating mutation responsive to targeted therapy (per NCCN guidelines)
5. No prior systemic therapy or radiotherapy for metastatic lung cancer (surgery alone permitted)
6. Planned treatment with targeted therapy specific to the oncogene driver mutation.
7. Declines repeat biopsy option or does not have tumor site amenable to biopsy.
8. Patients must have the ability to understand and willingness to sign an informed consent document.

Immunotherapy Cohort - Blood Draw Only

1. Have a histologically confirmed diagnosis of locally advanced or stage IV NSCLC without a treatable activating mutation that would be amenable to targeted therapy AND planned first line treatment with immunotherapy or chemotherapy plus immunotherapy.
2. Aged 18 years or older
3. ECOG 0-2
4. No prior systemic therapy or radiation therapy for lung cancer (surgery alone permitted)
5. Patients must have the ability to understand and willingness to sign an informed consent document.

Exclusion Criteria:

Targetable Oncogene - Biopsy Cohort (includes blood draw)

1. Concurrent health problem which would preclude tissue biopsy (e.g. hemophilia or other bleeding predisposition).
2. Patients whose only biopsy source would involve sampling an anatomic area that carries an unacceptably high procedural risk (e.g. pericardium or kidney) as deemed by the treating physician or by a proceduralist performing the biopsy.
3. Patients whose only biopsy source involves a sample that may not be evaluable due to insufficient genomic material (such as cerebrospinal or ascitic fluid) as deemed by the treating physician. .

Targetable Oncogene Cohort and Immunotherapy Cohort - Blood Draw Only

1. Planned follow up on therapy outside of the University of Colorado Health System
2. Unwillingness to allow for residual clinical biopsy specimens to be utilized in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have a diagnosis of State IV Lung Adenocarcinoma with EGFR activating mutation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05-10 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
gene expression changes | baseline and 2 weeks (+/- 1 week) for each patient.
  change from baseline of tumor gene expression profile at 2 weeks. Global gene expression data will be collected using RNAseq
protein expression change | baseline and 2 weeks (+/- 1 week) for each patient.
  change from baseline of protein gene expression profile at 2 weeks as measured by multiplex protein assay (proteins to be assayed include: e-cadherin, vimentin, fibronectin, CD4, CD8, CD14, CD16, CD206, PDL1, and CSF1R)

SECONDARY OUTCOMES:
Depth of Response | Study startup through 36 months
  Correlation between the depths of tumor response (by RECIST v1.1) (percentage decrease in tumor size) with the presence of an EMT signature.

OTHER OUTCOMES:
Evaluation of Adverse Events | Study startup through 36 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Success rate of Repeat Biopsy | Study startup through 36 months
  Success rate of early rebiopsy in obtaining tumor samples that have evaluable material for RNA Seq and other analyses
Progression Free Survival | Study startup through 36 months
  Length of PFS as per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Erin Schenk, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No